CLINICAL TRIAL: NCT01576562
Title: Implantable Cardioverter Defibrillator (ICD) Function During Ventricular Assist Device (VAD) Implantation
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM13674
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Heart Failure
Keywords: Implantable Cardioverter Defibrillator; Ventricular Assist Device
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group - Control Group: VAD implantation (study group) or other cardiothoracic surgery (control group)

SUMMARY:
The purpose of this research study is to test the function of a subjects implantable cardioverter defibrillator (ICD) function throughout the duration of their heart surgery. ICD function can be altered during some types of heart surgery such as those when a pump (ventricular assist device - VAD) is implanted. The investigators would like to study the mechanism of device and ICD malfunction.

DETAILED DESCRIPTION:
ICD function is typically measured prior to and after surgery. For the study, the investigators will measure ICD lead function multiple times throughout the surgery as well, to determine if and when device malfunction occurs. ICD lead function is measured noninvasively through a specialized computer the same way it is checked in the clinic. In addition, the investigators will test ICD function as they usually do following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18 and older
* Have a wireless implantable cardioverter defibrillator (ICD) and are undergoing VAD implantation or other cardiothoracic surgery.

Exclusion Criteria:

* Patients who are pacemaker dependent
* children, human fetuses, neonates
* prisoners will not be included
* Pregnant women will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with wireless ICDs undergoing VAD implantation (study group) or other cardiothoracic surgery (control group) will be included.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
observational study to assess potential changes that may occur in the RV ICD lead function during LVAD implantation and what mechanism may cause those changes in RV ICD lead function | RV ICD lead function will be measured throughout LVAD placement , at 1 week post LVAD placement, and 3 months post LVAD placement Description:

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Kron, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Hu YL, Kasirajan V, Tang DG, Shah KB, Koneru JN, Grizzard JD, Ellenbogen KA, Kron J. Prospective Evaluation of Implantable Cardioverter-Defibrillator Lead Function During and After Left Ventricular Assist Device Implantation. JACC Clin Electrophysiol. 2016 Jun;2(3):343-354. doi: 10.1016/j.jacep.2016.01.008. Epub 2016 Mar 23. PMID 29766894